CLINICAL TRIAL: NCT04205942
Title: Cold Plasma Therapy for Acceleration of Wound Healing in Superficial, Infected Diabetic Foot
Brief Title: Cold Plasma Therapy for Acceleration of Wound Healing in Diabetic Foot
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Diethelm Tschoepe, Prof. Dr. Dr. med., Medical Director Diabetes Center at Herz- und Diabeteszentrum NRW, Ruhr University of Bochum
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KPW2016-1.1
Record Dates: First submitted 2019-12-12; First posted 2019-12-20 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Diabetic Foot
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plasma (Experimental): regular treatment with Argon Plasma Jet according to manufacturer's instructions, 8 times within 14 days
  Interventions: Device: Argon Plasma Jet
- Placebo (Sham Comparator): Sham-treatment with Argon Plasma Jet, Plasma producing electric field switched off - no Plasma is produced, just argon gas as effluent, 8 times within 14 days
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Argon Plasma Jet — Cold Plasma (CP) therapy is applied in the first week of treatment on a daily schedule, in the second week CP is applied every second day. In total, 8 applications are performed with a one day schedule variance.
  Arms: Plasma
Device: Placebo — Sham Cold Plasma (sham-CP) (switched off Electric field, no plasma production, just gas) therapy is applied in the first week of treatment on a daily schedule, in the second week sham-CP is applied every second day. In total, 8 applications are performed with a one day schedule variance.
  Arms: Placebo

SUMMARY:
Diabetic foot is a common complication of diabetes mellitus and requires specialized treatment. Wounds are characterized by persistent infection and chronic inflammatory processes, impeding well directed matrix remodelling and wound closure. Cold plasma applications have demonstrated beneficial effects on wound healing in several case reports. The investigator-initiated "Kaltplasma Wund (KPW)-Trial" was performed to prove beneficial effects of cold plasma in wound healing in a prospective, placebo-controlled, randomized bi-center study.

DETAILED DESCRIPTION:
Diabetic foot (DF) is a major complication in patients with diabetes leading to increased risk of hospitalization, lower limb amputation, and death, as well as a significant decrease in quality of life. During lifetime the risk for developing DF is assumed to be 25%; with 30% of DF resulting in lower limb amputation. If compared to general population people with diabetes have a 20-fold higher risk for amputation. Diabetes mellitus is the leading cause of lower limb amputation. Ulceration and impaired wound healing are commonly associated with common co-morbidities; the increased risk of infection amongst patients with diabetes is driving chronification and accounts for lack of wound healing.

Non-thermal atmospheric pressure plasma has been proposed as a tool for various biological and medical applications relying on its capacity to reduce bacterial load in the wound and to initiate wound healing. Biological plasma effects are largely dependent on plasma-generated reactive species in the gas phase, which subsequently diffuse or react with proteins and lipids in cells or tissues.

Thus, the objective of this placebo-controlled patient-blinded study was to show that application of cold plasma in addition to standard care treatment compared to placebo could accelerate wound healing in terms of more rapid and clinical meaningful wound surface regression. Wound closure progression and microbiological analysis were monitored time dependently to prove the effects. Patient's well-being and subjective perceptions were evaluated during treatment.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or Type 2 Diabetes mellitus
* HbA1c ≤ 10%
* at least one chronic wound persisting for at least three weeks without healing tendency following standard care wound therapy (Armstrong Wagner Grade Ib or IIb)

Exclusion Criteria:

* concomitant wound treatment with local vacuum therapy or maggot therapy
* dialysis
* use of topical active antibiotics,
* concomitant treatment with platelet rich fibrin,
* presence of critical limb ischemia defined as ankle brachial index below 0.5 or transcutaneous oxygen pressure below 15 mmHg.
* participation in another clinical trial
* women of child bearing potential without effective contraception or active breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2016-08-17 (Actual); Primary Completion 2019-04-20 (Actual); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
change in wound surface area | treatment period of max 15 days
  change in wound surface area within 14 days treatment
change in signs of clinical infection | treatment period of max 15 days
  change in clinical signs of infections as judged by the investigator
change in microbial load | treatment period of max 15 days
  change in microbial count, being evaluated by microbial culture

SECONDARY OUTCOMES:
time to significant wound surface area change | treatment period of max 15 days
  time to 10% reduction of wound surface compared to treatment start
total wound surface change during treatment | treatment period of max 15 days
  total wound surface change compared to treatment start
time to change in wound infection | treatment period of max 15 days
  change in wound infection over treatment
changes in Quality of life (EQ5D questionnaire) | treatment period of max 15 days
  Evaluation of life quality during (EQ5D questionnaire) treatment period via questionaire
changes in Quality of life (SF12 questionnaire) | treatment period of max 15 days
  Evaluation of life quality during (SF12 questionnaire) treatment period via questionaire
treatment related side effects - formation of keloids | treatment period of max 15 days
  question to evaluate potential side effects of the therapy: formation of keloids will be answered in a "yes" or "no" fashion and reported
treatment related side effects - presence of skin irritation | treatment period of max 15 days
  question to evaluate potential side effects of the therapy: presence of skin irritation will be answered in a "yes" or "no" fashion and reported
treatment related side effects - local bleeding | treatment period of max 15 days
  question to evaluate potential side effects of the therapy: local bleeding will be answered in a "yes" or "no" fashion and reported
treatment related side effects - proliferative skin reaction | treatment period of max 15 days
  question to evaluate potential side effects of the therapy: proliferative skin reaction will be answered in a "yes" or "no" fashion and reported

OTHER OUTCOMES:
treatment related side effects - formation of keloids | within 5 years after start of treatment (at 1, 2 and 5 years after start of treatment)
  descriptive evaluation of side effects within 5 years after Treatment (at 1, 2 and 5 years after start of treatment) question to evaluate potential side effects of the treatment: formation of keloids will be answered in a "yes" or "no" fashion and reported
treatment related side effects - presence of skin irritation | within 5 years after start of treatment (at 1, 2 and 5 years after start of treatment)
  question to evaluate potential side effects of the therapy: presence of skin irritation will be answered in a "yes" or "no" fashion and reported
treatment related side effects - local bleeding | within 5 years after start of treatment (at 1, 2 and 5 years after start of treatment)
  question to evaluate potential side effects of the therapy: local bleeding will be answered in a "yes" or "no" fashion and reported
treatment related side effects - proliferative skin reaction | within 5 years after start of treatment (at 1, 2 and 5 years after start of treatment)
  question to evaluate potential side effects of the therapy: proliferative skin reaction will be answered in a "yes" or "no" fashion and reported

CONTACTS AND LOCATIONS:
Overall Officials: Diethelm Tschoepe, Prof, Principal Investigator — Herz- und Diabeteszentrum NRW, Ruhr-Universität Bochum

IPD SHARING:
Plan to Share IPD: No
no sharing of patient data planned, data are analysed locally

REFERENCES:
- [Derived] Hiller J, Stratmann B, Timm J, Costea TC, Tschoepe D. Enhanced growth factor expression in chronic diabetic wounds treated by cold atmospheric plasma. Diabet Med. 2022 Jun;39(6):e14787. doi: 10.1111/dme.14787. Epub 2022 Jan 21. PMID 35007358
- [Derived] Stratmann B, Costea TC, Nolte C, Hiller J, Schmidt J, Reindel J, Masur K, Motz W, Timm J, Kerner W, Tschoepe D. Effect of Cold Atmospheric Plasma Therapy vs Standard Therapy Placebo on Wound Healing in Patients With Diabetic Foot Ulcers: A Randomized Clinical Trial. JAMA Netw Open. 2020 Jul 1;3(7):e2010411. doi: 10.1001/jamanetworkopen.2020.10411. PMID 32672829